CLINICAL TRIAL: NCT05904392
Title: Effect of Music Therapy on the Anxiety Level of Patients During the Administration of Ocular Intravitreal Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Collaborators: University of Vic - Central University of Catalonia (Other)
Responsible Party: Principal Investigator, Eduard Pedemonte-Sarrias, MD, PhD, Althaia Xarxa Assistencial Universitària de Manresa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CEI 22/109
Record Dates: First submitted 2023-05-28; First posted 2023-06-15 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Anxiety and Fear
Keywords: Music therapy; anxiety; intravitreal injection; pain; quality of life
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Music played prior to intravitreal injection
  Interventions: Other: Music
- Control (No Intervention): No music played.

INTERVENTIONS:
Other: Music — Music played prior to injection
  Arms: Intervention

SUMMARY:
Introduction Ocular intravitreal injection is a widely used ophthalmic invasive technique to administer medication directly inside the patient's eye. Despite being usually a quick and painless intervention, some patients report nervousness and anxiety before and during the procedure. Music therapy could help in assessing this discomfort, as previous studies have shown it can beneficial, specially helping to reduce anxiety levels.

Objective This study aims to assess the effect of music therapy on patients undergoing intravitreal injections and how it affects their anxiety.

Methods This is a randomized, prospective, single blind, clinical trial. Patients will be divided into two groups. Group A patients will listen to classical music during the procedure (intervention). Group B patients (control), will not listen to music during the procedure. All other aspects of the procedure will be the same for both groups. To analyze the impact music therapy, patients will fill in the STAI anxiety questionnaire and will be evaluated with the pain visual analogue scale (VAS) before and after the injection procedure.

Expected results Subjects that undergo the procedure with music therapy are expected to experience less anxiety that the ones that do not. Less pain perception is also expected.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years old.
* Patients must have been prescribed an intravitreal injections of an anti-VEGF drug.
* Subjects must have undergone at least one previous intravitreal injection.
* Patients must fully understand the procedure and the project they will be participating in and agree on signing the informed consent.

Exclusion Criteria:

* Patients with a psychiatric diagnosis with the need to take anxiety medication.
* Patients that before the intervention took medication to relax, such as benzodiazepines or anxiolytics.
* Subjects with hearing difficulty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
STAI | Just before and immediately after intervention
  Change in anxiety score test

CONTACTS AND LOCATIONS:
Locations (1):
- Eduard Pedemonte Sarrias, Manresa, Barcelona, Spain